CLINICAL TRIAL: NCT00597545
Title: Effect of Augmentation of Cerebral Blood Flow on Neuropsychometric Performance After Carotid Endarterectomy in Type II Diabetic Patients
Brief Title: Effect of Raised CBF During CEA on Cognition in DM Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Half of DM patients had EEG changes and therefore were excluded.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eric J. Heyer, MD, PhD, Professor of Clinical, Department of Anethesiology Clinical Operations, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAC3837
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Carotid Artery Disease; Carotid Artery Stenosis; Diabetes; Cognitive Dysfunction
Keywords: Carotid Endarterectomy; Neuropsychological tests; Stroke; Transient ischemia; Hypoperfusion; Ischemia
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Diabetes Mellitus; Cognitive Dysfunction; Stroke; Ischemia | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Shunt (Active Comparator): Patients with diabetes mellitus (DM) undergoing carotid endarterectomy will receive a shunt only if it is indicated by EEG, by "conventional" management.
  Interventions: Procedure: Carotid endarterectomy; Device: Shunt
- Prophylactic Shunt (Experimental): Patients with diabetes mellitus (DM) undergoing carotid endarterectomy will receive a shunt even when by standard criteria they would not need to receive one.
  Interventions: Procedure: Carotid endarterectomy; Device: Shunt

INTERVENTIONS:
Procedure: Carotid endarterectomy — When a shunt is inserted to increase blood flow to the brain
Device: Shunt — A tube inserted below and above the surgical area at the time when the carotid artery is clamped to allow the surgeon to work in a bloodless field and to supplement blood flow to the brain.

SUMMARY:
The purpose of this study is to determine if we can reduce the incidence of cognitive dysfunction - difficulty in performing certain pencil-paper, memory, finger dexterity and thinking type of tasks called neuropsychometric tests - in patients with adult onset diabetes mellitus (DM) undergoing surgery on the carotid artery (CEA).

We hypothesize that cognitive dysfunction can be decreased in patients with type II DM by augmenting cerebral blood flow with a shunt during carotid endarterectomy compared to patients with Type II DM who are treated with "conventional" management in which a shunt is placed only if the electroencephalogram (EEG) indicates cerebral ischemia.

DETAILED DESCRIPTION:
Based on previous clinical studies, we have found that patients with diabetes mellitus (DM) who are having carotid endarterectomy (CEA) have a four-fold higher incidence of cognitive dysfunction, 1 day and 1 month after surgery, than a control group of elderly diabetic patients having spine surgery.

We hypothesize that this increased incidence is due to sub-cortical ischemia associated with the clamping of the ipsilateral carotid artery, because intra-operatively we rarely see EEG changes, or a significant number of emboli upon clamping or unclamping the carotid artery, or new cortical lesions of ischemia by MRI after surgery. In order to decrease cognitive dysfunction in patients with DM, we propose to randomize them to either i) have a shunt placed across the surgical site assuming it is surgically feasible or ii) be treated by "conventional" management during which time a shunt is placed only in the unlikely event of significant cortical ischemia determined by EEG, which occurs in about 5% of all cases.

The purpose of this study is to determine if patients with adult-onset diabetes mellitus having the surgical procedure called carotid endarterectomy benefit from increasing blood flow to the brain with a "shunt". A "shunt" is a tube inserted below and above the surgical area at the time when the carotid artery is clamped to allow the surgeon to work in a bloodless field and to supplement blood flow to the brain. Benefit is measured after surgery by comparing performance on a battery of cognitive tests, which test your ability to perform pencil-paper, memory and finger dexterity tests, to performance before surgery.

Patients in the shunt group whom the surgeon at the time of surgical exposure considers too technically difficult to shunt, will not have a shunt inserted but will be treated statistically as if they were shunted (intention to treat). Follow-up evaluations will be performed 1 day, and 1 and 6 months after surgery so that the long-term effect of shunting can be evaluated.

Cerebral injury will be determined in two ways.

First, all patients will be evaluated using a battery of neuropsychometric tests before and after surgery. Patients admitted to the Irving Clinical Research Center (CRC) will have their tests 1 day before, and 1 day, and 1 and 6 months after surgery. Those coming into the hospital on the day of surgery, "Same Day", will be evaluated on the day of surgery. They will be evaluated 1 day, and 1 and 6 months after surgery.

Preoperative neurological and neuropsychological evaluation will be performed. The neuropsychometric tests are not intended to be diagnostic of specific neuropsychiatric disorders, but rather are designed to demonstrate general neuropsychological pathology. These tests can be divided into four types: (1) an evaluation of language, (2) an evaluation of speed of mental processing, (3) an evaluation of ability to learn using a list of words, and (4) an evaluation of visual perception requiring a patient to copy a complex figure. Before the battery is administered we will assess each patient's level of pain while sitting and standing using a 10 point Visual Analog Scale and gauge their mood with a series called the Wong/Baker Faces Rating scale. Patients having spine surgery may have significant pain before surgery which might impair their performance.

We will also be measuring Quality of Life (QOL) in all enrolled patients.

This will be done using two well-known examinations (Telephone Interview for Cognitive Status (TICS) and Centers for Disease Control and Prevention Health-Related Quality-of-Life 14Item Measure (CDC HRQOL14)) and a series of questions investigating how well patients are able to perform activities of daily living (ADLs) and instrumental activities of daily living (IADLs). These tests will be given at two time points, once before the surgery and then one month after surgery. We will look for changes in quality of life that may correlate with neuropsychometric test performance.

Second, peripheral serum samples will be drawn before induction, before crossclamping the carotid artery, 15 minutes after crossclamping the carotid artery and 24 hours after surgery.

Since the purpose of this study is to determine if a change in "conventional" management will improve patient's ability to perform our battery of neuropsychometric tests, we will randomly assign patients to either receive a "shunt" prophylactically if the surgeon determines that it is technically safe, even if conventional management does not indicate its necessary, or a "shunt" only if it is indicated by EEG, "conventional" management. Subjects in the prophylactic group will receive a shunt even when by standard criteria they would not need to receive one. Randomization will be performed in blocks of four patients each using a randomization table. Using "block" randomization we will increase the probability of an equal number of patients "shunted" or not shunted. The surgeon will be told which group the patient has been randomized into after induction and prior to clamping the carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak English
* no history of permanent neurological impairment, Axis I psychiatric diagnosis or drug abuse
* scheduled for elective carotid endarterectomy for treatment of carotid artery stenosis
* diagnosed with diabetes mellitus or HbA1c value greater than 10%

Exclusion Criteria:

* younger than 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Heyer, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, Department of Anesthesiology, New York, New York, United States

REFERENCES:
- [Result] Heyer EJ, Mergeche JL, Bruce SS, Connolly ES. Inflammation and cognitive dysfunction in type 2 diabetic carotid endarterectomy patients. Diabetes Care. 2013 Oct;36(10):3283-6. doi: 10.2337/dc12-2507. Epub 2013 Jun 4. PMID 23735728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Shunt | Prophylactic Shunt
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Shunt | Prophylactic Shunt | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Full Range); unit: years] | 68 [64 to 78] | 69 [65 to 79] | 68.7 [64 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Neuropsychometric Changes
Description: Battery of neuropsychometric tests to evaluate a variety of cognitive functions.
Time Frame: Post-operatively at 1 day
Measure: Number; unit: participants
Arm/Group | Conventional Shunt | Prophylactic Shunt
Number analyzed (Participants) | 4 | 6
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 1 post-op
Arm/Group | Conventional Shunt | Prophylactic Shunt
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No